CLINICAL TRIAL: NCT05393193
Title: Point-of-Care HIV Testing and Early Dolutegravir Use for Infants
Brief Title: POC HIV Testing and Early DTG Use for Infants
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Botswana Harvard AIDS Institute Partnership (Other); Ragon Institute of MGH, MIT and Harvard (Other); Botswana Ministry of Health (Other Government); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Roger Shapiro, Associate Professor of Immunology and Infectious Diseases, Harvard School of Public Health (HSPH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 155BHP; P01HD107670 (NIH)
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIV-exposed neonates (Other): Point-of-care HIV testing at birth
  Interventions: Diagnostic Test: Point-of-Care Cepheid Xpert HIV-1
- HIV-positive infants identified through birth HIV screening (Other): Early antiretroviral treatment per standard of care, including dolutegravir-based regimen beginning at 4 weeks of age for infants weighing at least 3.0kg.
  Interventions: Drug: DTG/ABC/3TC

INTERVENTIONS:
Diagnostic Test: Point-of-Care Cepheid Xpert HIV-1 — Post-partum HIV-positive women with pre-determined risk factors for vertical HIV transmission will be offered point-of-care HIV testing for their newborns for early infant HIV diagnosis.
  Arms: HIV-exposed neonates
Drug: DTG/ABC/3TC — Infants will be started on a combination of NVP/ZDV/3TC. A switch to DTG/ABC/3TC will occur for all infants at or after 4 weeks (28 days) post-delivery for those weighing ≥3kg. Dosing of all ART will be weight-based by the Botswana treatment guidelines.
  Arms: HIV-positive infants identified through birth HIV screening

SUMMARY:
This study is being conducted to explore the feasibility of implementing targeted birth HIV testing of high-risk neonates using facility-based point-of-care (POC) HIV diagnostics, and to improve the ability to implement the best standard-of-care treatment possible. Infants found to be HIV infected will be immediately offered enrollment into a dolutegravir (DTG) antiretroviral treatment study cohort (if maternal consent is granted) or referred for treatment at a government facility. Infants who enter the study treatment cohort will be prospectively followed through 96 weeks of age. ART will follow Botswana guidelines.

ELIGIBILITY:
Inclusion criteria for point-of-care infant HIV testing:

1. Mother 18 years of age or older
2. Mother willing and able to provide verbal consent for infant testing
3. Infant birth weight ≥1.5kg
4. Presence of any of the following risk factors:

<12 weeks of ART prior to delivery (including no ART); Known HIV-1 viremia (above level of detection) for last test performed or at any time >24 weeks gestation in pregnancy; CD4 cell count known to be <350 cells/mm3 within the past year; Self-described poor adherence in pregnancy (1 or more complete days of missed ART)

Exclusion criteria for point-of-care infant HIV testing:

1) Medical condition making it unlikely that the infant will survive to 24 months

Inclusion criteria for infant longitudinal treatment cohort:

1. Mother 18 years of age or older
2. Mother willing and able to provide written informed consent for study participation for herself and her infant
3. Positive point-of-care HIV screening for infant (HIV DNA PCR pending or completed)
4. Infant eligible for ART treatment in accordance with the Botswana government program
5. Infant birth weight ≥1.5 kg

Exclusion criteria for infant longitudinal treatment cohort:

1. Medical condition making it unlikely that the infant will survive to 24 months
2. Infant unable to start treatment-dose ART < 168 hours of age
3. Infant unable to attend follow-up visits at a BHP study clinic in Gaborone or Francistown

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-07-04 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of high-risk HIV-exposed infants identified and tested | within 72 hours of life
  Analysis will largely be descriptive, highlighting the proportion of high-risk infants identified and tested at each facility. Proportions will be determined by populating actual numbers approached and screened matched against exact denominators obtained from surveillance data.
Median time to HIV diagnosis and treatment-dose ART | 7 days
  We will describe the proportion of high-risk infants found to be HIV positive per risk category and compare this to findings from another cohort study of early-treated children. Average time to HIV diagnosis and treatment initiation will also be described.
The proportion of children with HIV-1 RNA <40 copies/mL at 12 weeks on ART | 12 weeks on ART
  We will compare time to viral suppression and the proportion with complete HIV-1 RNA suppression (<40 copies/mL) at 12 weeks from ART start between infants on early DTG with another cohort of children on early LPV/r.
The proportion of children with successful DTG-based treatment through 96 weeks on ART | 96 weeks on ART
  We will compare the proportion with complete HIV-1 RNA suppression and no need for treatment modification at all visits through 96 weeks between infants on early DTG with another cohort of children on early LPV/r.
The proportion of infants with grade 3 or 4 adverse events/hospitalization/death | 96 weeks on ART
  We will compare the proportion with grade 3 or 4 adverse events through 96 weeks between infants on early DTG with another cohort of children on early LPV/r.

CONTACTS AND LOCATIONS:
Overall Officials: Roger L Shapiro, MD, MPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Botswana Harvard HIV/AIDS Institute Partnership, Gaborone, Botswana